CLINICAL TRIAL: NCT03867370
Title: A Phase Ib/II, Open-Label, Multi-Center Study Evaluating the Efficacy and Safety of Neoadjuvant Toripalimab Injection (JS001) or Toripalimab in Combination With Lenvatinib for Patients With Resectable Hepatocellular Carcinoma (HCC)
Brief Title: Toripalimab in Combination With Lenvatinib as Neoadjuvant Therapy in Resectable Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Enrollment is over, the study was completed
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JS001-020-Ib-HCC
Record Dates: First submitted 2019-03-01; First posted 2019-03-08 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — toripalimab; lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): During the neoadjuvant period, the patients will receive a single dose JS001 intravenous infusion of 480 mg. After the operation, the patients will receive JS001 240 mg Q3W for up to 48 weeks.
  Interventions: Drug: Toripalimab (JS001 )
- Group B (Toripalimab, Lenvatinib) (Experimental): During the neoadjuvant period, the patients will receive a single dose JS001 intravenous infusion of 480 mg in combination with oral lenvatinib at a starting dose of 8 or 12 mg once a day. After the operation, the patients will receive JS001 240 mg Q3W and lenvatinib for up to 48 weeks.
  Interventions: Drug: Toripalimab (JS001 ) Lenvatinib
- Group C (Toripalimab, Lenvatinib) (Active Comparator): During the neoadjuvant period, the patients will receive a single dose JS001 intravenous infusion of 480 mg in combination with oral lenvatinib at a starting dose of 8 or 12 mg once a day. After the operation, the patients will receive JS001 240 mg Q3W for up to 48 weeks.
  Interventions: Drug: Toripalimab (JS001 ) Lenvatinib

INTERVENTIONS:
Drug: Toripalimab (JS001 ) — Given IV
  Arms: Group A
Drug: Toripalimab (JS001 ) Lenvatinib — Given IV 4 mg capsules
  Arms: Group B (Toripalimab, Lenvatinib)
Drug: Toripalimab (JS001 ) Lenvatinib — Given IV 4 mg capsules
  Arms: Group C (Toripalimab, Lenvatinib)

SUMMARY:
This study will evaluate efficacy and safety of Toripalimab Injection (JS001) with or without Lenvatinib as a Neoadjuvant Therapy in patients with Resectable Hepatocellular Carcinoma (HCC)

ELIGIBILITY:
Confirmed by histopathological or cytological examination; The criteria for resectability is met; Has at least one evaluable lesion according to the RECIST 1.1 standard and has not received local treatment;

Exclusion Criteria:

Patients who previously received anti-programmed death receptor-1 (PD-1) antibody, anti-programmed death ligand-1 (PD-L1) antibody, anti-programmed death ligand-2 (PD-L2) antibody or anti-cytotoxic T lymphocyte-associated antigen-4 (CTLA-4) antibodies, including those who have participated in a JS001 clinical study;

Patients with a history of gastroesophageal varices or active cardia ulcers associated with a high risk of bleeding; Patients who have upper gastrointestinal hemorrhage within 1 year; Patients known to have fibrous layer HCC, sarcomatoid HCC or mixed cholangiocarcinoma and HCC; Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Pathological response rate | Up to 2 months
  CPR，MPR

SECONDARY OUTCOMES:
Objective response rate | up to 2 months
  ORR is defined as the percentage of participants who achieved CR or PR
Percentage of R0 resection | up to 8 months
  Used for assessment of the feasibility of the neoadjuvant therapy.
Time to operation | up to 8 months
  Used for assessment of the feasibility of the neoadjuvant therapy.
Progression free survival | up to 3 years
  Used for assessment of the efficacy.
Overall survival | up to 3 years
  Used for assessment of the efficacy.
Incidence of adverse events | up to 3 years
  Graded using the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Safety will be recorded through the incidence of adverse events, serious adverse events and specific laboratory abnormalities (worst grade) in each treatment arm.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Zhongshan Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Fang Y, Liu W, Tang Z, Ji X, Zhou Y, Song S, Tian M, Tao C, Huang R, Zhu G, Jiang X, Gao J, Qu W, Wang H, Zhou P, Wu X, Jin L, Sun H, Ding Z, Peng Y, Zhao S, Zhou J, Fan J, Xu W, Shi Y. Monocarboxylate transporter 4 inhibition potentiates hepatocellular carcinoma immunotherapy through enhancing T cell infiltration and immune attack. Hepatology. 2023 Jan 1;77(1):109-123. doi: 10.1002/hep.32348. Epub 2022 Feb 7. PMID 35043976